CLINICAL TRIAL: NCT00594334
Title: Effect of Actonel on Periodontal Health of Postmenopausal Women
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 010706
Expanded Access: Available
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Periodontal Disease
Keywords: osteopenia; periodontitis
MeSH Terms: conditions — Periodontal Diseases; Bone Diseases, Metabolic; Periodontitis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- E, I (Experimental)
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — Weekly Risedronate

SUMMARY:
Hypothesis: Women who use Actonel (risedronate) for osteopenia will show beneficial periodontal effects.

DETAILED DESCRIPTION:
Women who use Actonel for osteopenia will show beneficial attachment loss, alveolar bone height and morphology as compared to those who do not when oral hygiene is corrected for.

ELIGIBILITY:
Inclusion Criteria:

* Osteopenia
* Postmenopausal

Exclusion Criteria:

* Male
* Diabetes

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal alveolar bone changes | one year

SECONDARY OUTCOMES:
Periodontal attachment levels | one year

CONTACTS AND LOCATIONS:
Overall Officials: james liu, md, Principal Investigator — University Hospitals Cleveland Medical Center; leena palomo, dds msd, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Uhcmc, Cleveland, Ohio, United States